CLINICAL TRIAL: NCT04423887
Title: Effects of Creatine Supplementation in Addition to Resistance Exercise Training in Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FUI/CTR/2020/5
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Electric Stimulation Therapy; Musculoskeletal Manipulations; Creatine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator)
  Interventions: Other: Lower Extremity Resistance Exercise Training; Other: Home Exercise Plan; Device: Electrotherapy + Heating; Procedure: Joint Mobilization
- Creatine Supplementation (Experimental)
  Interventions: Other: Lower Extremity Resistance Exercise Training; Other: Home Exercise Plan; Device: Electrotherapy + Heating; Procedure: Joint Mobilization; Dietary Supplement: Creatine Supplementation

INTERVENTIONS:
Other: Lower Extremity Resistance Exercise Training — Treadmill walking 5-10 min for warm up Strength training: (80% of 8RM)
  3 times supervised exercise for 4 weeks Warm up (Self Paced walking for 10 minutes) leg press, leg extension, Sit to stand squat (mini squats) Stationary Cycling (Maximum Resistance as per patient tolerance till failure)
  3 sets 8 reps 10-15 s rep rest interval 1-2 min set rest interval
  Other Names: Lower Extremity Strength Training
Other: Home Exercise Plan — 2 sets of 10 repetitions/day of
  AROM isolated knee extension and knee flexion Isometric isolated knee extension and knee flexion Isometric terminal knee extension Sit to stand squat Isometric knee terminal extension
Device: Electrotherapy + Heating — Interferential Current therapy (2P), in combination with heating pad for 20 minutes
Procedure: Joint Mobilization — Tibio-femoral Anterior Glide Tibio-femoral Posterior Glide Patellofemoral Joint Mobilization
  Other Names: Manual Therapy
Dietary Supplement: Creatine Supplementation — Creatine Supplementation 20g/day for 1 week followed by 5 g/day for 3 weeks
  Arms: Creatine Supplementation

SUMMARY:
Despite the past decade being dedicated to bone and joint disease, the incidence and prevalence rates of osteoarthritis continues to rise, and till date not curative treatment has been identified for the management of knee osteoarthritis. In terms of conservative management of knee osteoarthritis, pharmacological management has been the mainstay of treatment, however is associated with numerous adverse effects with prolonged use, and it is important to look into the non-pharmacological alternates for the management of knee osteoarthritis. Research has shown resistance exercise training to be the most effective non-pharmacological treatment option for the management of knee osteoarthritis, and the purpose of the current study is to determine if the addition of a non-pharmacological dietry supplement like creatine can amplify the beneficial effects of resistance exercise training in patients with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-70 years
* Knee OA with history not less than three months.
* Radiological evidences of grade III or less on Kellgren classification.
* Knee pain on VNRS no more than 8/10

Exclusion Criteria:

* Neuromuscular conditions that may lead to fatigue such as multiple Sclerosis
* Signs of serious pathology (e.g., malignancy, inflammatory disorder, infection).
* History of trauma or fractures in lower extremity.
* Signs of lumbar radiculopathy or myelopathy.
* History of knee surgery or replacement.
* Patients on intra-articular steroid therapy within two months before the commencement of the study.
* Impaired skin sensation.
* Impaired renal function

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2020-12-06 (Actual); Study Completion 2020-12-06 (Actual)

PRIMARY OUTCOMES:
Knee Pain: Visual Analogue Scale | 2 weeks
  Visual Analogue Scale was used to measure pain scoring from 0-10 cm on a horizontal 10cm line. A greater score reflects higher pain intensity.
Knee Pain: Visual Analogue Scale | 4 weeks
  Visual Analogue Scale was used to measure pain scoring from 0-10 cm on a horizontal 10cm line. A greater score reflects higher pain intensity.
Knee Range of Motion | 2 weeks
  Knee Range of Motion will be quantified by using Gonimeter
Knee Range of Motion | 4 weeks
  Knee Range of Motion will be quantified by using Gonimeter
Knee Isometric Muscle Strength | 2 weeks
  Knee Isometric Muscle Strength will be quantified by using Modified Sphygmomanometer Dynamometer
Knee Isometric Muscle Strength | 4 weeks
  Knee Isometric Muscle Strength will be quantified by using Modified Sphygmomanometer Dynamometer
Six Minute Walk Test | 2 weeks
  Six Minute Walk Test will be used to quantify walking related performance fatigability, walking distance and walking speed.
Six Minute Walk Test | 4 weeks
  Six Minute Walk Test will be used to quantify walking related performance fatigability, walking distance and walking speed.
5 repetition sit to stand test | 2 weeks
  Time will be measured to perform 5 repetitions of sit to stand activity. Lesser time means a better score.
5 repetition sit to stand test | 4 weeks
  Time will be measured to perform 5 repetitions of sit to stand activity. Lesser time means a better score.

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) | 2 weeks
  Knee Injury and Osteoarthritis Outcome Score (KOOS) to measure physical function and quality of life. A greater score on Knee Injury and Osteoarthritis Outcome Score reflects good prognosis and outcome and a lower score shows poor prognosis and outcome. the score for Knee Injury and Osteoarthritis Outcome Score is reported in the form of percentage i.e. 0-100%.
Knee Injury and Osteoarthritis Outcome Score (KOOS) | 4 weeks
  Knee Injury and Osteoarthritis Outcome Score (KOOS) to measure physical function and quality of life. A greater score on Knee Injury and Osteoarthritis Outcome Score reflects good prognosis and outcome and a lower score shows poor prognosis and outcome. the score for Knee Injury and Osteoarthritis Outcome Score is reported in the form of percentage i.e. 0-100%.
Body Composition | 2 weeks
  Body Composition was measured via bioelectrical impedance analysis. A greater Phase angle reflects better cellular integrity and smaller phase angle reflects poorer cellular integrity.
Body Composition | 4 weeks
  Body Composition was measured via bioelectrical impedance analysis. A greater Phase angle reflects better cellular integrity and smaller phase angle reflects poorer cellular integrity.
Fall Risk | 2 weeks
  Fall risk will be quantified by using Biodex balance System
Fall Risk | 4 weeks
  Fall risk will be quantified by using Biodex balance System

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Osama, PhD*, Principal Investigator — Foundation University Institute of Rehabilitation Sciences
Locations (1):
- Foundation University Institute of Rehabilitation Sciences, Islamabad, Federal, Pakistan